CLINICAL TRIAL: NCT03323255
Title: Influence of the Modulation of the Posterior Parietal Cortex (rTMS) on a Pointing Movement With the Paretic Upper Limb After Stroke
Brief Title: rTMS Posterior Parietal Cortex Modulation and Upper Limb Movement After Stroke
Acronym: PPCstim
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016_36; 2016-A01608-43 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-10-16; First posted 2017-10-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Stroke; Hemiparesis; Transcranial Magnetic Stimulation; Brain Connectivity
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cTBS stimulation (Active Comparator): continuous theta-burst TMS stimulation (1200 pulses, 50Hz, separated in two sequences of 600 pulses)
  Interventions: Device: repeated transcranial magnetic stimulation continuous theta-burst stimulation
- SHAM stimulation (placebo) (Sham Comparator): SHAM stimulation
  Interventions: Device: SHAM repeated transcranial magnetic stimulation

INTERVENTIONS:
Device: repeated transcranial magnetic stimulation continuous theta-burst stimulation — cTBS
  Arms: cTBS stimulation
Device: SHAM repeated transcranial magnetic stimulation — SHAM stimulation
  Arms: SHAM stimulation (placebo)

SUMMARY:
This study evaluates the effect of a unique session of inhibitory rTMS (cTBS) over the contralesional posterio parietal cortex (PPC) on the spatio-temporal parameters of a pointing movement performed by stroke patients with their paretic upper limb. It will also assess the effects on the resting motor threshold of both hemispheres and on parietopremotor connectivity.

To achieve theses aims, the real cTBS stimulation will be randomly counterbalanced with a SHAM stimulation (in a second session) in a crossover design. Assessments will be performed before and after each stimulation session.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80y
* Right-handed
* Right hemispheric stroke confirmed by a 3D imaging technique
* at the chronic phase (>6months)
* subject being able to perform a pointing movement of at least 20cm in the anterior space without compensatory movements of the trunk
* informed consent
* Social security affiliation

Exclusion Criteria:

* Severe comprehension troubles (language, cognitive or psychiatric disorders)
* History of neurological disorders in addition to the stroke
* Locomotor troubles affecting the paretic arm
* Contraindication to rTMS : epilepsy, intracranial metallic foreign body, cochlear implant, unstable fracture of the skull bones, deafness
* pregnancy or breastfeeding
* adult subject to guardianship

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Time of movement during the pointing movement | 30 minutes
  Time between the initiation of the movement and the reaching of the target

SECONDARY OUTCOMES:
Reaction time (time between the go signal and th onset of the movement) | 30 minutes
  temporal parameters of pointing movements
Response time (time between the go signal and the reaching of the target) | 30 minutes
  temporal parameters of pointing movements
Peak velocity of the hand during the pointing movement | 30 minutes
  pak velocity in m/s
smoothness (number of units of movement during the pointing movement), | 30 minutes
  Spatial parameters of pointing movements
Linearity (ration between the length of the trajectory of the hand and the linear distance between the initial position of the hand and the target) | 30 minutes
  Spatial parameters of pointing movements
Detection of mirror movements with the healthy upper limb | 30 minutes
  EMG detection
Primary motor cortex excitability of both motor cortices | 30 minutes
  Resting motor threshold of lesioned and non-lesioned hemispheres
Parietomotor connectivity in the contralesional hemisphere | 30 minutes
  Assessed by a paired-pulse TMS protocol (see Allart et al. 2017 for more details)
Spatial bias | 30 minutes
  Line bisection test

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Allart, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Swynghedauw, CHU lille, Lille, France

IPD SHARING:
Plan to Share IPD: No